CLINICAL TRIAL: NCT01151072
Title: A Trial Comparing the Pharmacokinetic and Pharmacodynamic Properties of NN1250 After Different Routes of Administration in Healthy Subjects
Brief Title: A Trial Comparing the Effect of NN1250 After Different Routes of Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-1992; 2009-017217-30 (EudraCT Number); U1111-1113-6783 (Other: WHO)
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- IDeg i.m. thigh (Experimental)
  Interventions: Drug: insulin degludec
- IDeg i.v. (Experimental)
  Interventions: Drug: insulin degludec
- IDeg s.c. abdomen (Experimental)
  Interventions: Drug: insulin degludec
- IDeg s.c. deltoid (Experimental)
  Interventions: Drug: insulin degludec
- IDeg s.c. thigh (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Each subject was randomly allocated to five single dose administrations of NN1250 subcutaneously (under the skin) in the thigh, the abdomen (stomach) and the deltoid (shoulder), intramuscularly (into the muscle) in the thigh and intravenously (into the vein), respectively, on five separate dosing visits.

SUMMARY:
This trial was conducted in Europe. The aim of this clinical trial was to compare the exposure and effect of NN1250 (insulin degludec) after different routes of injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history, physical examination, vital signs and ECG (electrocardiogram), as judged by the Investigator
* Body mass index 18.0-27.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Area under the serum Insulin Degludec concentration-time curve (only for subcutaneous administration) | From 0 to 120 hours after single-dose

SECONDARY OUTCOMES:
Area under the serum Insulin Degludec concentration-time curve (only for intramuscular administration) | From 0 to 120 hours after single-dose
Area under the serum Insulin Degludec concentration-time curve (only for intravenous administration) | From 0 to 30 hours after single-dose
Maximum observed serum Insulin Degludec concentration after single-dose (only for subcutaneous and intramuscular administration) | Within 0 to 120 hours after dosing
Back-extrapolated initial serum Insulin Degludec concentration after single-dose (only for intravenous administration) | At time zero after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Nosek L, Coester HV, Roepstorff C, Thomsen HF, Kristensen NR, Haahr H, Heise T. Glucose-lowering effect of insulin degludec is independent of subcutaneous injection region. Clin Drug Investig. 2014 Sep;34(9):673-9. doi: 10.1007/s40261-014-0218-x. PMID 25124362
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com